CLINICAL TRIAL: NCT04825951
Title: Three Dimensional Evaluation Of Dentofacial Effects Of Two Non-Compliance Appliances In The Treatment Of Growing Skeletal Class III Patients (A Randomized Controlled Clinical Trial)
Brief Title: Dentofacial Effects Of Two Non-Compliance Appliances In The Treatment Of Growing Skeletal Class III Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Bassant Alaa, principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 070320212
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Malocclusion, Angle Class III
Keywords: Cone beam computed tomography; growing skeletal Class III; CS 2000® appliance; Reversed Forsus Fatigue resistant device
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial, parallel design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and statistician will be blinded (double blind) to the intervention group. After data collection is completed, the randomization code will be broken to reveal the allocation group. The operator will be blinded during recording of the measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CS 2000 appliance (Active Comparator): treating growing skeletal Class III patients
  Interventions: Other: CS 2000
- Reversed Forsus Fatigue resistant appliance (Active Comparator): treating growing skeletal Class III patients
  Interventions: Other: CS 2000
- Control (No Intervention): A group of untreated skeletally growing class III patients will be recruited to account for the possible effects of growth in the treatment groups.
  This group matches the treated groups in malocclusion, stages of skeletal maturation, and mean observation period. Those patients will be treated after the period of the study.

INTERVENTIONS:
Other: CS 2000 — treating growing Skeletal growing Class III patients
  Other Names: Reversed Forsus Fatigue resistant appliance
  Arms: CS 2000 appliance; Reversed Forsus Fatigue resistant appliance

SUMMARY:
Early orthodontic treatment of Class III malocclusions with skeletal and dentoalveolar imbalances, represents a continuous dilemma. This difficulty starts from their meticulous diagnosis and treatment planning till reaching satisfactory results and finally stability. Some appliances could be used to correct growing skeletal Class III patients, improving the skeletal and dentoalveolar relationships, creating proper conditions for final orthodontic treatment, more importantly avoiding surgery. These appliances remove patient compliance from the equation.

DETAILED DESCRIPTION:
Aim of the work: Evaluate the skeletal, dentoalveolar and soft tissue effects of two different force application systems which are the pulling force (CS 2000® appliance/ CS appliance) and the pushing force (Reversed Forsus fatigue-resistant device/ RF appliance).

Materials and methods: A randomized controlled clinical trial will be conducted to address the aim of the study. Thirty three growing skeletal Class III patients (9-11 years) will be recruited upon a lateral cephalometric x-ray. Subjects complying with the inclusion criteria will be randomly assigned using a computer-generated list to one of the three groups Group I: Eleven patients treated with CS2000 appliance, Group II: Eleven patients treated with reversed Forsus Fatigue Resistant device and Group III: control group of Eleven untreated patients with a ratio of 1:1:1 allocation. A CBCT will be made before installing the appliances. After gaining a 2 mm positive overjet or a 6 months period, alginate impressions will be poured and dental casts will be made. Photographs and CBCTs will also be performed to record the dentofacial effect of the used appliances.

Keywords: Cone beam computed tomography, growing skeletal Class III, CS 2000® appliance, Reversed Forsus Fatigue resistant device.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 8 years to 11 years.
* Cervical vertebrae maturation index (CVMI 2 and 3) identified on the lateral cephalometric radiograph.
* Angle Class III molar relation.
* Skeletal class III ANB ranges between (-4) - (0).
* Wits appraisal ranges between (0) - (-5).
* Patients with good oral hygiene, and a healthy periodontal condition.
* Reversed over jet (-1) - (-6).
* Normal vertical growth pattern (SN/MP angle 28˚-38˚).

Exclusion Criteria:

* A discrepancy between centric relation and maximum intercuspation.
* Patients who underwent previous orthodontic treatment.
* Patients currently receiving drug therapy that may affect orthodontic tooth movement.
* Congenitally missing teeth or extracted teeth.
* History of systemic disease or craniofacial syndromes or presence of cleft.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Skeletal readings angles | 6 months
  SNA in degrees SNB in degrees ANB in degrees SN-MP in degrees
Skeletal readings percetanges | 6 months
  LAFH in percentage
Skeletal readings in millimeters | 6 months
  Wits appraisal in millimeters
Dental readings angles | 6 months
  U1-PP in degrees U1- NA in degrees L1-MP in degrees L1-NB in degrees
Dental readings in millimeters | 6 months
  U1-NA millimeters L1-NB in millimeters.
Soft tissue readings in millimeters | 6 months
  UL- E plane in millimeters LL- E plane in millimeters

SECONDARY OUTCOMES:
Changes in airway | 6 months
  difference in airway volume in cubic millimeters .
Changes in TMJ | 6 months
  anterior, posterior, superior and medial joint space in cubic milimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant A Abbas, PHD resident, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
TREATMENT OF GROWING SKELETAL CLASS III PATIENTS

REFERENCES:
- [Background] Oliveira PM, Cheib-Vilefort PL, de Parsia Gontijo H, Melgaco CA, Franchi L, McNamara JA Jr, Souki BQ. Three-dimensional changes of the upper airway in patients with Class II malocclusion treated with the Herbst appliance: A cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2020 Feb;157(2):205-211. doi: 10.1016/j.ajodo.2019.03.021. PMID 32005472
- [Result] World Medical Association.. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. Bull World Health Organ. 2001;79(4):373-4. Epub 2003 Jul 2. No abstract available. PMID 11357217